CLINICAL TRIAL: NCT04646421
Title: Responsible Gambling Telephone Intervention to High-risk Gamblers by a State-owned Gambling Operator in Sweden. Effectiveness, User Satisfaction and Acceptability of the Motivational Telephone Intervention of AB Svenska Spel.
Brief Title: Responsible Gambling Telephone Intervention to High-risk Gamblers by a State-owned Gambling Operator in Sweden.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Collaborators: AB Svenska Spel (Unknown)
Responsible Party: Sponsor
Other Study IDs: omsorgssamtal
Record Dates: First submitted 2020-11-06; First posted 2020-11-30 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Problem Gambling; Gambling Disorder
Keywords: problem gambling; gambling disorder; behavioral addiction; motivational intervention; COVID-19
MeSH Terms: conditions — Gambling; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Motivational intervention - clients reached: Gamblers successfully reached with the motivational telephone intervention.
  Interventions: Behavioral: Motivational telephone intervention
- Control group: clients not reached for the motivational intervention: Clients aimed to be reached for the same intervention, but who were not reached and therefore were not exposed to the intervention.
- Prospective intervention group: Clients subject to the prospective study part (target N 200), who are successfully reached by the intervention from November, 2020, and who provide informed consent to the web survey study. Studied as a cohort without control group, but with the pre-intervention situation as their own control condition.
  Interventions: Behavioral: Motivational telephone intervention

INTERVENTIONS:
Behavioral: Motivational telephone intervention — Motivational telephone intervention to high-risk gamblers, aiming to stimulate them to reduce gambling, quit gambling, or to seek peer support or treatment.
  Groups: Motivational intervention - clients reached; Prospective intervention group

SUMMARY:
The present overall project evaluates an intervention carried out by the Swedish state-owned gambling operator AB Svenska Spel, in order to help high-risk gamblers reduce or quit their gambling. The intervention is a motivational telephone intervention, called by responsible gambling officers trained in motivational interviewing, and who call gamblers who are screened for suspected high-risk gambling practices either through the operator's own records, or because they have voluntarily taken a self-test indicating a hazardous gambling pattern. The present projects evaluates the effectiveness, user satisfaction and acceptability of the intervention, in two parts: 1) A retrospective, register-based follow-up of gamblers reached by the telephone intervention, in comparison to control individuals for whom attempts were made to carry out the same intervention, but who were never successfully reached on telephone. The effectiveness measures include potential changes in gambling level (frequency, level of wagering) post-intervention compared to pre-intervention, as well as occurrence of deposit limits, or voluntary self-exclusion. 2) A prospective web survey study involving individuals reached with the intervention from November, 2020, who - after receiving electronic written information and after providing informed consent - will answer a web survey around 10 days after the intervention, about their attitudes to the telephone intervention, and their self-reported gambling (on the same operator and on other gambling operators), self-limiting interventions and treatment seeking after the intervention. The study will provide important data on the effectiveness of this intervention aiming to reduce high-risk gambling practices, and will be able to study also the risk of gamblers transferring their gambling practices to other operators after a motivational intervention as the present one. Also, as acceptability and user satisfaction of the intervention are crucial for its success over time, these measures are also included in order to improve the understanding or how effective responsible gambling interventions can be implemented by gambling operators with a harm-reducing mission.

DETAILED DESCRIPTION:
The project includes two sub-studies:

1. Retrospective study part: intervention group (reached with the telephone intervention) and control group (gamblers attempted to be reached but who were not reached by the telephone intervention). Involves objective gambling data post- and pre-intervention, as derived from the AB Svenska Spel databases. Includes the study period September, 2019-April, 2020. Total N of individuals available: 3,626.

   This study part will also include a sub-analysis, where each individual successfully reached for the motivational telephone call will be compared to a 1:1-matched individual who was not reached (but intended to be reached by the call). Matching is carried out based on the reason for including the individual in the intervention, i.e. either because of a risk screen in a voluntary self-test, or the level of monthly gambling loss. An individual will be matched to a control individual based on the 2,000-SEK interval (approximately 190-Euro inteval) of gambling losses or the inclusion criterion of self-test risk screen.
2. Prospective study part: cohort study of individuals reached with the intervention prospectively from November, 2020, and who provide informed consent. Web survey study which collects data on user satisfaction, acceptability, and self-reported changes in gambling (on the same gambling operator and other gambling operators) post-intervention compared to self-reported gambling prior to the intervention. Data collected after sending the survey on the first business day 10 days after the intervention. Target N 200.

The aims of the study are the following:

1. Retrospective study part: to study 1a) effects of the telephone intervention, with respect to individuals' level of gambling (frequency and total amount), uptake of responsible gambling tools, and enrolment into self-exclusion, during four weeks after the intervention, in comparison to a period of eight weeks prior to the intervention; 1b) whether the objective effects above differed during the period of COVID-19 pandemic in Sweden (week by week throughout March and April, 2020, compared to previous weeks during the study)
2. Prospective study part: to study 2a) participants' subjective attitudes to and experience of the telephone intervention 2b) subjective effects of the intervention on participants' self-reported change in gambling on the same and other operators, and self-reported uptake of self-exclusion

ELIGIBILITY:
Inclusion Criteria:

* High-risk gambler as perceived by the high-risk gambling screen by the gambling operator (AB Svenska Spel) or by a voluntary self-test

Exclusion Criteria:

* None in the retrospective study. In the prospective study: failure to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who are gamblers and the AB Svenska Spel sub-section for sports and casino gambling, and who are screened as high-risk gamblers based on an objective measure from the operator or by a voluntary self-test taken by the gambler and indicating a high-risk gambling behavior.
  Study population retrospective study part: All individuals aimed for the telephone intervention September, 2019-April, 2020, comparing those who were successfully reached by the intervention, to the control individuals (not reached on telephone),
  Study population prospective study part: Individuals who are reached by the telephone intervention from prospective study start I November, 2020, and who receive a text message intervention 10+ days after the intervention (first business day 10 days after the intervention) and who provide informed consent to study participation.
Sampling Method: Non-Probability Sample
Enrollment: 3626 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in gambling frequency. | 4 weeks
  Change in wagering (any, and frequency) for each of the specific gambling types, during four weeks after the intervention, compared to the eight weeks prior to the intervention.
Change in money wagered | 4 weeks
  Change in wagering (amounts) for each of the specific gambling types, during four weeks after the intervention, compared to the eight weeks prior to the intervention.
Change in money lost | 4 weeks
  Change in losses for each of the specific gambling types, during four weeks after the intervention, compared to the eight weeks prior to the intervention.
Occurrence of any self-limiting intervention post-intervention | 4 weeks
  Occurrence of deposit limits and voluntary self-exclusions post-intervention,during four weeks after the intervention, compared to the eight weeks prior to the intervention.
Change in wagering frequency in both the own operator and other operators | 10 days
  Reduced wagering frequency for each of the specific gambling types, during the approximate 10-day period after the intervention, in gamblers reached with the intervention in the prospective study part (self-reported in survey sent on first business day 10 days after the intervention)
Change in wagering amounts in both the own operator and other operators | 10 days
  Reduced wagering (amounts) and losses for each of the specific gambling types, during the approximate 10-day period after the intervention, in gamblers reached with the intervention in the prospective study part (self-report in survey sent on first business day 10 days after the intervention)
Change in gambling losses in both the own operator and other operators, in prospective study part | 10 days
  Gambling losses (amounts) for each of the specific gambling types, during the approximate 10-day period after the intervention, in gamblers reached with the intervention in the prospective study part (survey sent on first business day 10 days after the intervention)
Occurrence of any self-limiting intervention after the intervention in prospective study part | 10 days
  Occurrence of self-reported voluntary self-exclusions and help-seeking during the approximate 10-day period after the intervention in the prospective study part (self-reported in survey sent on first business day 10 days after the intervention)

SECONDARY OUTCOMES:
Gambler's immediate perception of the call | 0 days
  Gambler's self-reported satisfaction (overall) with the call, as responded by telephone to a direct question from the caller, in the retrospective study part
Gambler's perception of the intervention | 10 days
  Gambler's attitudes to positive and negative effects of the call (feelings of care from the operator and feelings or being annoyed by the call), in the prospective study part (survey sent on first business day 10 days after the intervention)
Gambler's perception of the intervention's effects on gambling | 10 days
  Gambler's attitudes to the call with respect to subjective effects on gambling (increasing/decreasing) and help-seeking, in the prospective study part.(survey sent on first business day 10 days after the intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No